CLINICAL TRIAL: NCT03887676
Title: A Randomized Placebo-controlled Trial of ARBaclofen vs. Placebo in the Treatment of Children and Adolescents With ASD
Brief Title: Arbaclofen vs. Placebo in the Treatment of Children and Adolescents With ASD (ARBA)
Acronym: ARBA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: McMaster University (Other); Western University, Canada (Other); Queen's University (Other); Unity Health Toronto (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARB-05-2018
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — arbaclofen placarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arbaclofen (Active Comparator)
  Interventions: Drug: Arbaclofen
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Arbaclofen — Administered orally as disintegrating tabs, round, white and beveled edges, at the following strengths: 5mg, 10mg, 15mg and 20mg
  Arms: Arbaclofen
Other: Placebo — Administered orally as disintegrating tabs, round, white and beveled edges
  Arms: Placebo

SUMMARY:
This study will examine the safety and efficacy of arbaclofen vs. placebo on social function in children and adolescents with Autism Spectrum Disorder (ASD).

DETAILED DESCRIPTION:
There are no pharmacologic treatments available for social function deficits in individuals with ASD. The data for pharmacologic treatment of repetitive behaviours in this disorder has also become difficult to interpret given that the last two large multisite trials of selective serotonin reuptake inhibitors (SSRIs) in autism are reported to be negative for the treatment of repetitive behaviours. Only the associated symptom of irritability has 2 drugs with Food and Drug Administration (FDA) indications, whereas no systematic data exists on the pharmacologic treatment of anxiety in ASD, and response to rates to stimulants for hyperactivity are lower than what is seen in Attention Deficit Hyperactivity Disorder (ADHD). In addition, there are no biological markers of treatment response identified in this population at this point. This study will examine the potential efficacy and safety of arbaclofen for social function, and will explore biological markers of safety and treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients 5-17 years of age inclusive.
2. Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). DSM-5 criteria will be established by a clinician with expertise with individuals with ASD. Diagnosis will be supported by the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2).
3. Complex language to qualify for ADOS-2 modules 3 or 4.
4. If already receiving stable concomitant medications affecting behaviour, have stable regimens with no changes during the preceding 6 weeks prior to Screening, and will not electively initiate new or modify ongoing medications for the duration of the study.
5. If already receiving stable non-pharmacological educational and behavioural interventions, have continuous participation during the preceding 3 months prior to Screening, and will not electively initiate new or modify ongoing interventions for the duration of the study.
6. Have normal physical examination and laboratory test results at Screening. If abnormal, the finding(s) must be deemed clinically insignificant by the Investigator.
7. Ability to obtain written informed consent from the participant, if developmentally appropriate. If a participant does not have the capacity to consent, ability to obtain assent (if developmentally appropriate), as well as written informed consent from their parent(s)/legal guardian(s).

Exclusion Criteria:

1. Pregnant females; sexually active females on inadequate birth control.
2. Have a serious medical condition that, based on Investigator judgment, might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. Have evidence of any significant hematological, endocrine, cardiovascular (including uncorrected symptomatic congenital heart disease), respiratory, renal, hepatic, or gastrointestinal disease, not including mild common pediatric diseases in these areas that are stable (e.g. mild asthma, constipation, etc.).
3. Have unstable epilepsy (i.e. seizures occurring within the last 6 months), or have epilepsy and not on stable doses of antiepileptic medications (i.e. dose changes within the last 3 months).
4. Have a history of drug abuse.
5. Have hypersensitivity to arbaclofen or any components of its formulation.
6. Unable to tolerate venipuncture procedures for blood sampling.
7. Actively enrolled in another intervention study.
8. Taking racemic bacblofen, vigabatrin, tiagapine, riluzole, clobazam or regular benzodiazepine use (prn and hs use is allowed).
9. Unable to take oral medications.
10. Known hypersensitivity to racemic baclofen.
11. Inability to speak and understand English sufficiently enough to allow for the completion of all study assessments (parent/legal guardian; participant).

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) - Social Domain | 16 weeks
  To examine the effect of arbaclofen vs. placebo social function

SECONDARY OUTCOMES:
Clinical Global Impressions - Impression Scale - Improvement (CGI-I) | 16 weeks
  To examine the effect of arbaclofen vs. placebo on measures of global function
Aberrant Behavior Checklist (ABC) - Social Withdrawal Subscale | 16 weeks
  To examine the effect of arbaclofen vs. placebo on social withdrawal
Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) - Communication Domain | 16 weeks
  To examine the effect of arbaclofen vs. placebo on communication
Safety Monitoring Uniform Report Form (SMURF) | 16 weeks
  To examine the safety and tolerability of arbaclofen in children and adolescents with ASD
Clinical Global Impressions - Impression Scale - Global (CGI-I-Global) | 16 weeks
  To examine the safety and tolerability of arbaclofen in children and adolescents with ASD
Epworth Sleepiness Scale for Children and Adolescents (ESS-CHAD) | 16 weeks
  To examine the safety and tolerability of arbaclofen in children and adolescents with ASD
Suicidality assessment using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 16 weeks
  To examine the safety and tolerability of arbaclofen in children and adolescents with ASD

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, M.D, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Robert Nicolson, M.D, Principal Investigator — University of Western Ontario, Lawson Health Research Institute; Julia Frei, M.D, Principal Investigator — McMaster University, Offord Centre for Child Studies; Muhammad Ayub, M.D, Principal Investigator — Queen's University
Locations (4):
- Canada (4):
  - McMaster University, Offord Centre for Child Studies, Hamilton, Ontario
  - Queen's Universtiy, Kingston, Ontario
  - University of Western Ontario, Lawson Health Research Institute, London, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711